CLINICAL TRIAL: NCT07348510
Title: Comparison Between the Diuretic Effect of Aminophylline and Furosemide in Adult Patients Undergoing Cardiac Surgical Procedures: A Randomized Controlled Trial
Brief Title: Diuretic Effect of Aminophylline and Furosemide in Adult Patients Undergoing Cardiac Surgical Procedures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Hassan, Assistant Lecturer of Anesthesia, surgical ICU and Pain management, Cairo University, Cairo, Egypt, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MD-258-2024
Record Dates: First submitted 2026-01-07; First posted 2026-01-16 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Diuretic Effect; Aminophylline; Furosemide; Cardiac Surgical Procedures
MeSH Terms: interventions — Aminophylline; Furosemide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aminophylline group (control group) (Active Comparator): Patients will receive Aminophylline.
  Interventions: Drug: Aminophylline
- Furosemide group (Experimental): Patients will receive furosemide.
  Interventions: Drug: Furosemide

INTERVENTIONS:
Drug: Aminophylline — Patients will receive Aminophylline.
  Arms: Aminophylline group (control group)
Drug: Furosemide — Patients will receive furosemide.
  Arms: Furosemide group

SUMMARY:
This work aims to investigate the diuretic effect of Aminophylline in comparison to Furosemide in adult patients undergoing cardiac surgical procedures.

DETAILED DESCRIPTION:
Acute Kidney injury (AKI) is a serious and common complication after either adult or pediatric cardiac surgery.

The results of a recent meta-analysis suggested that loop diuretics (furosemide) may reduce postoperative creatinine clearance, whereas aldosterone agonists (spironolactone) increase the incidence of cardiac surgery-associated acute kidney injury (CSA-AKI). Diuretics are not recommended for the prevention of AKI, but loop diuretics may be used for the management of volume overload Aminophylline in cardiac surgery can reduce the frequency of AKI and could be used in the prevention of AKI as a safe and efficient modality in high-risk patients.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18-65 years.
* Both sexes.
* All adult patients presenting for elective cardiac surgical procedures performed on cardiopulmonary bypass (Coronary artery bypass surgery, Cardiac valve repair and/or replacement, Repair of large septal defects, Repair and/or palliation of congenital heart defects, Transplantation, surgery of thoracic aneurysms.).
* Body mass index (BMI) ranged between 20 and 40 kg/m2.

Exclusion Criteria:

* Sensitivity or contraindication to Aminophylline or furosemide
* Stage-5 chronic kidney disease (CKD) [Glomerular filtration rate (GFR) of less than 15 mL/min].
* The presence of both factors (GFR less than 60 mL/min and albumin greater than 30 mg per gram of creatinine) along with abnormalities of kidney structure or function for greater than three months signifies chronic kidney disease.
* Recipients of dialysis before surgery.
* Recipients of solid-organ transplantation before surgery.
* Emergency cardiac surgical procedures (e.g. left main coronary artery bypass graft, stuck valves, etc).
* Patient refusal.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2026-01-17 (Actual); Primary Completion 2026-07-26 (Estimated); Study Completion 2026-07-26 (Estimated)

PRIMARY OUTCOMES:
Measurement of urine output | Two hours after cardiopulmonary bypass
  Urine output will be measured at two hours after cardiopulmonary bypass.

SECONDARY OUTCOMES:
Measurement of urine output at completion of cardiopulmonary bypass | 48 hours after cardiopulmonary bypass
  Urine output at completion of cardiopulmonary bypass (CPB) will be measured at 8 hours and 48 hours after CPB.
Urea level | 48 hours after cardiopulmonary bypass
  Urea level will be measured at 8 hours and 48 hours after cardiopulmonary bypass.
Creatinine level | 48 hours after cardiopulmonary bypass
  Creatinine level will be measured at 8 hours and 48 hours after cardiopulmonary bypass.
Lactate level | 48 hours after cardiopulmonary bypass
  Lactate level will be measured at 8 hours and 48 hours after cardiopulmonary bypass.
Estimated Glomerular Filtration Rate (eGFR) | 48 hours after cardiopulmonary bypass
  Estimated Glomerular Filtration Rate (eGFR) at completion of cardiopulmonary bypass (CPB) will be measured at 8 hours and 48 hours after CPB.
Measurement of fluid balance | 48 hours after cardiopulmonary bypass
  Fluid balance at completion of cardiopulmonary bypass (CPB) will be measured at 8 hours and 48 hours after CPB.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.